CLINICAL TRIAL: NCT02323230
Title: Phase 2 Study of an Immunotherapeutic Vaccine, DPX-Survivac With Low Dose Cyclophosphamide in Patients With Recurrent Survivin-Expressing Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Study of DPX-Survivac Vaccine Therapy in Patients With Recurrent Survivin-expressing DLBCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: new study
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-DPX-Survivac-05
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2018-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DPX-Survivac + low dose cyclophosphamide (Experimental)
  Interventions: Biological: DPX-Survivac; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: DPX-Survivac — Immunotherapeutic vaccine targeting survivin antigen will be administered subcutaneously
Drug: Cyclophosphamide — Low dose cyclophosphamide will be taken by mouth

SUMMARY:
This phase 2 study was designed to assess the efficacy and safety of DPX-Survivac plus low dose cyclophosphamide in up to 24 subjects with recurrent diffuse large B-cell lymphoma (DLBCL) who are not eligible for transplant. However, with the evolving field of immunotherapy Immunovaccine has begun to focus on combination therapies, combining DPX-Survivac treatment with checkpoint inhibitors and other immune modulators. This phase 2 study was therefore terminated with fewer subjects than planned to allow the progress of other studies, such as NCT03349450.

DETAILED DESCRIPTION:
A multi-center treatment study assessing the efficacy and safety of an immunotherapeutic vaccine (DPX-Survivac) combined with low dose cyclophosphamide. Subjects with measurable, histologically proven DLBCL expressing survivin will be treated in this open-label, single arm study. Survivin is a protein commonly over-expressed in many types of cancer, including DLBCL.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects with histologically proven recurrent DLBCL. Subjects may have recurrence after primary or second treatment regimens for DLBCL. Subjects with recurrence at least 90 days post-autologous stem cell transplantation (ASCT) are eligible. Patients with partial response or measurable disease after first line therapy (who are not candidates for ASCT) or after second line therapy without disease progression may also be eligible.
* Previous localized surgery, radiotherapy, and chemotherapy more than 21 days prior to SD0.
* Subjects may have received previous courses of an investigational biologic therapy including active or passive immunotherapy (e.g. rituximab), other B cell depleting antibody therapy, or radioimmunotherapy (e.g. tositumomab or ibritumomab) if last administration is greater than 77 days prior to SD0.
* Subjects must have at least one measurable site of disease.
* Willing to undergo a pre-treatment and post-treatment tumor biopsy.
* Subjects must have evidence of survivin expression in pre-treatment tumor sample.
* A screening Eastern Cooperative Oncology Group Performance Status (ECOG) of 0-1.
* A life expectancy > 6 months.

Main Exclusion Criteria:

* Patients eligible for possible curative therapies such as ASCT.
* Patients undergoing concurrent chemotherapy, radiation therapy, or immunotherapy or who are currently on an investigational product/trial are excluded. There must be at least 21 days since completion of prior chemotherapy/radiation and at least 77 days since completion of immunotherapy until study treatment begins (SD0). Subjects must have recovered from all acute toxicities from prior treatment; peripheral neuropathy must be < grade 2.
* Lactate dehydrogenase (LDH) greater than 2 times the upper limit of normal.
* Patients with refractory disease after their last treatment (i.e. progression within 90 days).
* Patients who have received prior survivin based vaccines.
* Progressive CNS lymphoma requiring treatment within 84 days prior to SD0.
* History of active autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis requiring treatment within the last two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate | approximately 6 months

SECONDARY OUTCOMES:
Immune response | 1 year
  levels of cell mediated immunity targeting the survivin epitopes
Frequency of adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario